CLINICAL TRIAL: NCT01362101
Title: Effect of Behavioral Training on Physiological Responses to Smoking Cues, Affect and Cortisol
Acronym: physio
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: A. Eden Evins (Other)
Responsible Party: Sponsor-Investigator, A. Eden Evins, Director Center for Addiction Medicine, Massachusetts General Hospital
Organization: Massachusetts General Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 2010P-001316
Record Dates: First submitted 2011-05-23; First posted 2011-05-27 (Estimated); Last update posted 2013-07-11 (Estimated); Status verified 2013-07

CONDITIONS: Smokers
Keywords: cue reactivity; physiologic activation; craving; smoking cues; Behavioral therapy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Traditional behavioral intervention (Active Comparator)
  Interventions: Behavioral: Mindfulness behavioral intervention (MT),cognitive behavioral intervention (CBT)
- Mindfulness behavioral intervention (Active Comparator)
  Interventions: Behavioral: Mindfulness behavioral intervention (MT),cognitive behavioral intervention (CBT)

INTERVENTIONS:
Behavioral: Mindfulness behavioral intervention (MT),cognitive behavioral intervention (CBT) — 60 smokers will enter a separate 4 wk group sessions trial that evaluates efficacy of MT in comparison to CBT for smoking cessation. During the parent study, participants will receive bi-weekly sessions of either MT or CBT, for 4 weeks and to set a quit date at the end of the 2nd week. In this context, we will examine participants at two points:
  * Week 0-1 of MT/CBT: development of smoking scripts based participant's descriptions of situations that trigger tobacco craving.
  * Then participants will undergo pre-treatment (week 0-1) and post treatment (week 4) psychophysiological activation to smoking-related cues using the script driven imagery technique, in vivo cues, salivary cortisol testing and to complete a computerized SST protocol.

SUMMARY:
This study is ancillary. Participants will be recruited as part of a separate clinical trial on effects of two intensive behavioral training programs that evaluates feasibility and efficacy of a behavioral treatment that includes mindfulness techniques (MT) in comparison to traditional behavioral therapy (CBT) for smoking cessation. The investigators propose to compare the effect of MT to that of traditional CBT on a physiological marker of stress, salivary cortisol concentration, and physiological responses to smoking cues in tobacco smokers. The investigators will use electrophysiological reactivity to smoking cues in the form of audio recordings of personalized scripts describing the scenarios associated with the strongest urges to smoke that will provide a physiological validation to a behavioral intervention. The investigators will also explore correlations between these biological markers and self report of stress, craving and negative affect to supplement self report and behavioral outcome measures with biological and physiological markers to represent improvement attributed to the intervention.

ELIGIBILITY:
Inclusion Criteria:

1. Inclusion Criteria for the entire trial:

   * Women and men aged 18-65, inclusive, who are competent, wish to participate and willing to provide informed consent.
   * Self report smoking >=15 cigarettes/day.
   * Expired air CO > 9ppm at the time of enrollment.
   * Must be willing to participate in a meditation training group.
2. Inclusion criteria for the physiological assessment:

   * Abstinent for at least 12 hrs prior to the assessment.
   * CO<15ppm
   * Have negative urine toxicology for illicit drugs or alcohol.

Exclusion Criteria:

* DSM-IV diagnosis of dementia, neurodegenerative disease, or other organic mental disorder, lifetime history of psychotic disorder, bipolar disorder, severe PTSD, Dissociative Identity Disorder, OCD, anorexia nervosa, mental retardation, or autism.
* History of moderate or severe major depressive episode or generalized anxiety disorder within the last 6 months.
* Use of prescribed psychotropic medication other than SSRI/NDRI/SNRI/ buprenorphine in past 6mo, or change in such psychiatric medication dose in past six months.
* History of active substance use disorder other than nicotine or caffeine in the last 6 months.
* Positive urine toxicology for illicit drugs, alcohol, opiates or benzodiazepines.
* Serious unstable medical illness including, cardiovascular, hepatic, renal, respiratory, endocrine, neurological, or hematological disease such that hospitalization for treatment of that illness is likely within the next 4 months. History of life-threatening arrhythmia, CHF, syncope, or myocardial infarction within the last year. Abnormal cardiovascular event, or uncontrolled hypertension within last 2 months.
* History of cerebro-vascular events (i.e., stroke, TIA), multiple head injuries with neurological sequelae, a single severe head injury with lasting neurological sequelae, history of seizure disorder or current CNS tumor.
* Use of investigational medication in the past 30 days.
* Inability to speak, read, or understand English.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2010-07; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
physiologic reactivity (skin conductance, Heart rate, electromyogram, cortisol measures) to smoking cues in recently abstinent tobacco smokers | It will be measured twice during the study: before treatment (baseline at week 0) and an average of 7 days after treatment (end point assessment)
  * Wk 0: development of scripts based on participant's descriptions of the most salient aspects of the smoking experience that triggers craving. Then they will undergo pre-treatment psychophysiological activation to smoking-related cues using the script driven imagery technique (smoking-related and affectively neutral scripts), in vivo cues and salivary cortisol testing.
  * Wk 4: After the last MT or CBT session, participants will undergo post-treatment psychophysiological activation to smoking-related cues using the script driven imagery technique, in vivo cues and salivary cortisol testing.

SECONDARY OUTCOMES:
self reported of cue-induced negative affect, craving, and stress in recently abstinent tobacco smokers | It will be measured twice at the baseline assessment (before and after script driven imagery) and twice at the end point assessment (before and after script driven imagery)

CONTACTS AND LOCATIONS:
Overall Officials: Gladys N Pachas, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Center For Addiction Medicine-Massachusetts General Hospital, Boston, Massachusetts, United States